CLINICAL TRIAL: NCT01708226
Title: Attention Training for Childhood Obsessive Compulsive Disorder: An Open Case Series
Acronym: AMPOCD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Susanna Chang, PhD, Assistant Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB12-001459; 1R34MH095885-01A1 (NIH)
Record Dates: First submitted 2012-10-11; First posted 2012-10-16 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Obsessive Compulsive Disorder
Keywords: OCD; obsessive compulsive disorder; children
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Adenosine Monophosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Attention Modification Program (Experimental): Attention Modification Program
  Interventions: Behavioral: Attention Modification Program

INTERVENTIONS:
Behavioral: Attention Modification Program — Computer-based attention training treatment designed to directly but implicitly modify biased attention patterns in anxious patients in service of symptom relief.
  Other Names: AMP

SUMMARY:
Pediatric Obsessive Compulsive Disorder (OCD) is a chronic, impairing condition that accrues significant concurrent and long-term risk to affected youth. Although empirically supported psychosocial and pharmacological treatments for OCD exist, many children and their families are not able to adequately access these treatments or derive only partial benefit from them. Such findings highlight the importance of developing more effective treatment options which have the potential to be widely accessible to OCD youth.

The investigators are proposing to test a computerized attention modification program, AMP, in six youth with OCD in an open case series to gather information regarding protocol acceptability, feasibility and preliminary efficacy. This phase includes the development and refinement of stimuli selection procedures, behavior avoidance task, EEG protocol, and AMP parameters for use with children.

Following ascertainment of study eligibility, participants will undergo a baseline assessment consisting of a clinical interview, neurocognitive assessments, EEG, attention bias assessment, and self report questionnaires. Study participants will then receive 12 sessions of AMP treatment over the course of three weeks. All youngsters and their families will be reassessed at treatment endpoint (week 4). Participation will take a total of about 24 hours over the course of six weeks. Participants who are treatment responders may be asked to return approximately 3 months after completing treatment for a follow-up assessment.

Preliminary hypotheses: 1) AMP will be acceptable to youth and families and feasible to administer; 2) Youth receiving AMP will demonstrate decreases in threat bias and OCD symptom severity.

ELIGIBILITY:
Inclusion Criteria:

* Youth ages 8 - 17
* Primary DSM-IV diagnosis of OCD as determined by Anxiety Disorders Interview Schedule (ADIS-IV) Child/Parent version
* Child Yale-Brown Obsessive Compulsive Scale (CYBOCS) score > 15
* Medication free or on stable medication for six weeks prior to study entry
* Informed parental consent and child assent. Parents must agree to their child's participation in this protocol. Parents will be asked to fill out self-report questionnaires and participate in assessments that will provide us with more information about their child, however parents are not considered "participants" within this protocol, as all treatment is targeted toward their child.

Exclusion Criteria:

* DSM-IV depressive disorder, bipolar disorder, PTSD, substance abuse/dependence, conduct disorder, PDD, schizophrenia, or mental retardation
* Concurrent psychosocial treatment for OCD
* IQ < 80
* Youngsters with other comorbid disorders (e.g., anxiety, ADHD, ODD, tic disorder) will be eligible as long as these disorders are secondary to OCD in terms of severity and impairment and do not require immediate treatment initiation.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2012-11; Primary Completion 2013-11 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Children's Yale-Brown Obsessive Compulsive Scale Change From Pre-Treatment to Post-Treatment | pre-treatment (week 0) and post-treatment (week 5)

SECONDARY OUTCOMES:
Clinical Global Impression-Severity (CGI-S) and Improvement (CGI-I) Scales Change From Pre-Treatment to Post-Treatment | pre-treatment (week 0) and post-treatment (week 5)
Attention Bias Assessment Change from Pre-Treatment to Post-Treatment | pre-treatment (week 0) and post-treatment (week 5)
  Computerized assessment of attention bias

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Chang, PhD, Principal Investigator — University of California, Los Angeles; John Piacentini, PhD, Principal Investigator — University of California, Los Angeles; James McCraken, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No